CLINICAL TRIAL: NCT03958916
Title: Prospective Multicenters Clinical Cohort Study on Efficacy and Safety of Stratified Treatment for Chinese Children With Burkitt Lymphoma/Diffuse Large B-cell Lymphoma
Brief Title: Prospective Multicenters Clinical Cohort Study of Stratified Treatment of Chinese Children With BL/DLBCL
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Xiao-Fei Sun, professor, Sun Yat-sen University
Other Study IDs: SCCCG-BL/DLBCL-2017-001
Record Dates: First submitted 2019-05-20; First posted 2019-05-22 (Actual); Last update posted 2022-05-09 (Actual); Status verified 2022-05

CONDITIONS: Rituximab; Lymphoma, Non-Hodgkin; Pediatric Cancer
MeSH Terms: conditions — Lymphoma, Non-Hodgkin; Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The trial SCCCG-BL/DLBCL-2017 is a collaborative prospective, multicenters, non-randomized, observational, cohort clinical study with participating centers of the South China Children's Cancer Group-Non-Hodgkin lymphoma group(SCCCG-NHL). The aim of the study is to evaluate efficacy and safety of stratified treatment based on risk factors of childhood and adolescents Burkitt lymphoma(BL)/diffuse large B-cell lymphoma(DLBCL) patients in china.

DETAILED DESCRIPTION:
Research purposes:

1. To investigate the efficacy and safety of SCCCG-BL/DLBCL-2017 in children with BL and DLBCL.
2. To investigate the effect of rituximab combined with chemotherapy on the survival rate of children with high-risk BL/DLBCL.
3. To investigate the effect of rituximab on immune function in children with high-risk BL/DLBCL.
4. To explore the correlation between MRD detection and the efficacy and survival of children with BL/DLBCL.
5. To explore the role of PET/CT in evaluating residual lesions in children after BL/DLBCL treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Age < 18 years old
2. Pathologically confirmed Burkitt lymphoma or diffuse large B-cell lymphoma
3. Newly diagnosed patients
4. Informed consent of guardian of children patients

Exclusion Criteria:

1. Pathological components with follicular lymphoma
2. Immunodeficiency Second neoplasm

Ages: 1 Year to 18 Years | Sex: All
Age Groups: Child, Adult
Study Population: Burkitt lymphoma/diffuse large B-cell lymphoma patients，age at diagnosis < 18 years.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2017-05-05 (Actual); Primary Completion 2022-05-05 (Estimated); Study Completion 2025-05-05 (Estimated)

PRIMARY OUTCOMES:
Event-free survival (EFS) | through study completion, maximal eight years
  EFS is defined as time from start of treatment/randomization up to event or to date of last contact for patients without event. The following occurrences are defined as an event: non-response, progressive disease or relapse, treatment related death, death of any other cause or diagnosis of secondary malignancies.
Immune reconstitution rate (only in intermediate/high risk patients | 12 months after start of treatment
  Immune reconstitution rate is defined as percentage of patients achieving age adjusted serum immunoglobulin levels 12 months after start of treatment.

SECONDARY OUTCOMES:
Overall survival (OS) | through study completion, maximal eight years
  OS is defined as time from start of treatment/randomization up to death of any
Relapse-free survival (RFS) | through study completion, maximal eight years
  RFS is defined as time from start of treatment/randomization up to event or to date of last contact for patients without event. The following occurrences are defined as an event: non-response, progressive disease, or relapse.
Response rate (RR) | on an average 3 weeks after finish of treatment
  Complete response, partial remission, objective effect, stable disease or progressive disease
Adverse event rate | from the first day of protocol defined treatment until two years after start of protocol defined treatment
  Rate of patients with acute toxicity defined as grade III/IV/V AE
Rate of patients achieving normal immunoglobulin level 12 months after start of treatment | 12 months after start of treatment
  Rate of patients achieving normal immunoglobulin level 12 months after start of treatment
Time interval to normal immunoglobulin level | through study completion, maximal eight years
  Time interval to normal immunoglobulin level

CONTACTS AND LOCATIONS:
Overall Officials: Sun Xiaofei, Master, Principal Investigator — Sun Yat-sen University
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Rosolen A, Perkins SL, Pinkerton CR, Guillerman RP, Sandlund JT, Patte C, Reiter A, Cairo MS. Revised International Pediatric Non-Hodgkin Lymphoma Staging System. J Clin Oncol. 2015 Jun 20;33(18):2112-8. doi: 10.1200/JCO.2014.59.7203. Epub 2015 May 4. PMID 25940716
- [Result] Bakhshi S, Radhakrishnan V, Sharma P, Kumar R, Thulkar S, Vishnubhatla S, Dhawan D, Malhotra A. Pediatric nonlymphoblastic non-Hodgkin lymphoma: baseline, interim, and posttreatment PET/CT versus contrast-enhanced CT for evaluation--a prospective study. Radiology. 2012 Mar;262(3):956-68. doi: 10.1148/radiol.11110936. PMID 22357895
- [Result] Goldman S, Smith L, Anderson JR, Perkins S, Harrison L, Geyer MB, Gross TG, Weinstein H, Bergeron S, Shiramizu B, Sanger W, Barth M, Zhi J, Cairo MS. Rituximab and FAB/LMB 96 chemotherapy in children with Stage III/IV B-cell non-Hodgkin lymphoma: a Children's Oncology Group report. Leukemia. 2013 Apr;27(5):1174-7. doi: 10.1038/leu.2012.255. Epub 2012 Sep 3. No abstract available. PMID 22940833
- [Result] Meinhardt A, Burkhardt B, Zimmermann M, Borkhardt A, Kontny U, Klingebiel T, Berthold F, Janka-Schaub G, Klein C, Kabickova E, Klapper W, Attarbaschi A, Schrappe M, Reiter A; Berlin-Frankfurt-Munster group. Phase II window study on rituximab in newly diagnosed pediatric mature B-cell non-Hodgkin's lymphoma and Burkitt leukemia. J Clin Oncol. 2010 Jul 1;28(19):3115-21. doi: 10.1200/JCO.2009.26.6791. Epub 2010 Jun 1. PMID 20516455